CLINICAL TRIAL: NCT02005757
Title: Open Label, Multicenter, Randomized Study to Assess the Efficacy and Safety of Mizoribine in Active Rheumatoid Arthritis Patients Unsuccessfully Treated With Disease-modifying Antirheumatic Drug
Brief Title: Efficacy and Safety Study of Mizoribine in Active Rheumatoid (AMOLED)
Acronym: AMOLED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32RA13007
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; RA; Mizoribine; DAS28; European League Against Rheumatism
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mizoribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bredinin tablet 150mg (Experimental): dosage form: Tablet, dosage: 150mg qd, Duration: for 6months
  Interventions: Drug: Bredinin tablet 150mg
- Bredinin tablet 50mg (Active Comparator): dosage form: Tablet, dosage: 50mg tid, Duration: for 6months
  Interventions: Drug: Bredinin tablet 50mg

INTERVENTIONS:
Drug: Bredinin tablet 150mg — Bredinin 150mg qd vs Bredinin 50mg tid
  Other Names: Mizoribine
  Arms: Bredinin tablet 150mg
Drug: Bredinin tablet 50mg — Bredinin 150mg qd vs Bredinin 50mg tid
  Other Names: Mizoribine
  Arms: Bredinin tablet 50mg

SUMMARY:
The purpose of this study is to access the efficacy and safety of Mizoribine 150mg qid and 50mg tid in active rheumatoid arthritis patients unsuccessfully treated with disease-modifying antirheumatic drug.

DETAILED DESCRIPTION:
1. EULAR Response after 24weeks of treatment
2. EULAR Response after 12weeks of treatment
3. DAS28 value change
4. KHAQ-20 value change

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 20 to 80 years old
* Signed and dated informed consent document indicating that the patient
* Patients must have a diagnosis of Rheumatoid Arthritis(RA) of at least 3months duration as defined by the 2010 American College of Rheumatology(ACR) Classification criteria.
* Patients should have a Disease Activity Score 28 greater than or equal to 3.2 (DAS28 ≥ 3.2) and have received treatment with more than 1 kind of disease-modifying antirheumatic drug(including MTX).
* ESR≥28mm/h or CRP≥1.0mg/dl at screening.

Exclusion Criteria

* At screening, patients have laboratory result as defined by : white blood cell ≤ 3,000/mm3

  , Hemoglobin < 8.5 g/dL, Platelet count < 100,000/mm3, Serum creatinine > 2.0 mg/dL, Aspartic Acid Transaminase/Alanine Transaminase ≥ 2*upper limit of normal , Uric acid ≥ 1.5*upper limit of normal
* Patient must not have bleeding disorder or taking anticoagulant. (But, lt is allowed to take 100mg/day of Asprin)
* Patients with a history of operation on index knee joint which could have influence on the result and need to have surgery as determined by investigator.
* Patients have severe infection, including moderate respiratory disease and have received treatment with systemic antibiotics within 2 weeks.
* Patients have cardiovascular disease or associated disease which is not controlled.
* Patients have a history of malignancy within 5years. (But, basal cell or squamous cell carcinoma or carcinoma in situ of the uterine cervix have been treated is allowed)
* Patients have hypersensitivity reaction on this drug.
* Patients on any other clinical trial or experimental treatment in the past 3months.
* Female patients who are breast feeding, pregnant or plan to become pregnant during the trial or for two months following study termination.
* Not allowable medication recorded below ; Intra-articular injections within weeks at baseline visit, Patients taking oral steroid over 10mg /day or using new treatment or changing dosage within 4weeks at baseline visit, Using new nonsteroidal antiinflammatory drug within 4 weeks or changing nonsteroidal antiinflammatory drug dosage within 2 weeks at baseline visit.
* Having experience of use biologic agent, immunosuppressant, cytostatic preparations within 8weeks at baseline visit. (But, Rituximab is not allowed within 6months)
* Start to treatment new disease-modifying antirheumatic drug or need to change dosage of disease-modifying antirheumatic drug which is taking on the trial. (Leflunomide(ARAVA®) is not allowed within 12weeks, But, Cholestyramine is allowed after 48 hours later stopping. if it use three times a day, 8g, for 11days)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two years

CONTACTS AND LOCATIONS:
Overall Officials: Sung Su Kim, M.D., Ph.D, Study Chair — Gangneng asan Medical center
Locations (7):
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang
  - Hallym University chuncheon Sacred Heart Hospital, Chuncheon
  - Eulji University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Kangwon National University Hospital, Kangwon
  - Kyung Hee University hospital, Seoul
  - Soon Chun Hyang University Hospital, Seoul